CLINICAL TRIAL: NCT01614301
Title: A Prospective Phase I and Consecutive Phase II, Two-arm, Randomized Multi-center Trial of Temsirolimus in Combination With Pioglitazone, Etoricoxib and Metronomic Low-dose Trofosfamide Versus Dacarbazine (DTIC) in Patients With Advanced Melanoma
Brief Title: Phase I and Consecutive Phase II, Two-arm, Randomized Multi-center Trial in Patients With Advanced Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Principal Investigator, Albrecht Reichle, Professor MD, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEL001
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Advanced Melanoma
Keywords: advanced Melanoma
MeSH Terms: interventions — Dacarbazine; trofosfamide; Etoricoxib; Pioglitazone; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm (Experimental): Temsirolimus: 15 or 25 mg iv weekly , week 1+.In the phase I part of the study the finally used dosis will be determined. Pioglitazone (Actos) 60 mg p.o. daily, day 1+. Etoricoxib (Arcoxia) 60 mg p.o. daily, day 1+ Trofosfamide (Ixoten) 50 mg p.o. thrice daily as metronomic angiostatically and immunomodulatory acting therapy, day 1+. Treatment until disease progression or toxicity
  Interventions: Drug: dacarbazine (DTIC), Trofosfamide, Etoricoxib, Pioglitazone, Temsirolimus
- Controll Arm (Other): Dacarbazine (DTIC) 1000 mg/m2 day 1, every 3 weeks. The total number of DTIC cycles should not exceed 6 cycles due to cumulative toxicity.
  Interventions: Drug: dacarbazine (DTIC), Trofosfamide, Etoricoxib, Pioglitazone, Temsirolimus

INTERVENTIONS:
Drug: dacarbazine (DTIC), Trofosfamide, Etoricoxib, Pioglitazone, Temsirolimus — Dacarbazine (DTIC) 1000 mg/m2 day 1, every 3 weeks The total number of DTIC cycles should not exceed 6 cycles due to cumulative toxicity.
  Temsirolimus: 15 or 25 mg iv weekly , week 1+.In the phase I part of the study the finally used dosis will be determined. Pioglitazone (Actos) 60 mg p.o. daily, day 1+. Etoricoxib (Arcoxia) 60 mg p.o. daily, day 1+. Trofosfamide (Ixoten) 50 mg p.o. thrice daily as metronomic angiostatically and immunomodulatory actingtherapy, day 1+. Treatment until disease progression or toxicity

SUMMARY:
A prospective phase I and consecutive phase II, twoarm, randomized multi-center trial of temsirolimus in combination with pioglitazone, etoricoxib and metronomic low-dose trofosfamide versus dacarbazine (DTIC) in patients with advanced melanoma

Phase I: To determine the dose of temsirolimus to be used in phase II part of the study

Phase II:

To determine overall survival Secondary objectives

* To evalulate response rate
* To evaluate time to progression (TTP)
* To evalulate time to partial response (time to PR or better)(TPR)
* To evaluate quality of life
* To evaluate tolerability and safety

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Must be histologically diagnosed with metastatic melanoma and LDH level > 0.8 ULN
* Measurable lesions
* Subjects must receive study medication as first-line therapy. Preceeding adjuvant therapies are allowed.
* BRAF V600 mutation analysis
* Sufficient bone marrow function: neutrophils ≥ 2x109/l, hemoglobin ≥10 g/dl, platelets ≥ 100x109/l
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 (see Post Text Supplement 3).
* Required laboratory results:

  1. Liver function: Total bilirubin < 1.5 times of upper limit of local institution (ULN), SGPT, SGOT ≤ 2.5 times of upper limit of local institution
  2. Renal function: serum creatinine ≤ 1.5 ULN
  3. PT-INR/PT <1.5 ULN
* Normal cardiac function
* Patients with prior thrombembolic event with adequate anticoagulation
* Life expectancy at least 3 months
* Written informed consent of the patient prior to screening procedures
* Patient must be available for treatment and follow-up
* Adequate contraception in women capable of bearing children and men with partner capable of bearing children (combined oral contraceptives, hormonereleasing intrauterine contraceptive device, hormonal contraceptive implants, hormonal contraceptive injectables, surgical sterilization)
* Any previous surgery must have taken place more than 4 weeks prior to inclusion
* Previous radiation therapy must have involved less than 25% of bone marrow, and must have been completed more than 4 weeks prior to inclusion.
* For patients with controlled diabetes mellitus glucose levels have to be monitored continuously and the treating diabetologist has to be informed about the study participation of the patient.
* Patients with wild-type BRAF

Exclusion Criteria:

* Documented brain metastases unless the patient has completed successful local therapy for central nervous system metastases and has been off of corticosteroids for at least 4 weeks before enrollment.
* Patients who require vitamin K antagonists except for low dose
* Patients with bladder cancer or bladder cancer in their medical history, patients with risk factors for bladder cancer (such as exposure to aromatic amines or heavy tobacco smokers), or macrohematuria of unknown origin
* Prior history of stroke
* Known hypersensitivity to study drugs or to any of the excipients
* Active infection > grade 2 NCI-CTC version 4.0
* Known diagnosis of HIV, hepatitis B, or hepatitis C infection.
* Severe, unstable, or uncontrolled medical disease which would confound diagnoses or evaluations required by the protocol, including cardiac insufficiency (NYHA I -IV) uncontrolled diabetes including diabetic ketoacidosis, chronic hepatic or renal disease, active uncontrolled infection and chronic inflammatory intestinal disease, autoimmune diseases, peripheral arterial disease, verified coronary heart disease, cerebrovascular disease, acute peptic ulcer or acute gastro-intestinal bleeding.
* Prior radiation therapy > 25% of bone marrow
* Regular blood transfusions
* Treatment with other experimental substances within 30 days before study start
* Prior immunotherapy with ipilimumab, vaccination, B-raf inhibitor
* Participation in another clinical trial within 30 days before study start or during the trial
* Unwilling or unable to comply with the protocol
* Pregnant or breastfeeding patients. Women of childbearing potential must have a negative pregnancy test performed 7 days prior start of treatment.
* Patients with seizure disorders requiring medication (such as steroids or antiepileptics)
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Major surgery within 4 weeks prior to start of study or incomplete wound healing
* Drug or alcohol abuse
* Psychological or social conditions that may interfere with the patients participation in the study or evaluation of the study results.
* Known (at time of entry) gastrointestinal disorder, including malabsorbtion or active gastric ulcer, present to the extent that it might interfere with oral intake and absorption of study medication
* Patients undergoing dialysis or creatinine clearance <30 mL per minute, defined according to MDRD
* Patients with medically uncontrolled hypertension (RR continuously > 140/90 mm Hg)
* Any previous or concurrent malignancy or any cancer unless curatively treated > 3 years prior to study entry except cervical carcinoma in situ or adequate basal cell carcinoma
* Any urothelial cell carcinoma in the medical history
* Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic type reactions after acetylsalicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors
* Patients with BRAF V600 mutant metastatic melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
response rate | 2014

SECONDARY OUTCOMES:
Time to progession | 2014

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Reichle, Professor, Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg, Regensburg, Bavaria, Germany